CLINICAL TRIAL: NCT05439382
Title: Very Long-term Analysis of Root Coverage Stability Using Subepithelial Connective Tissue Graft Techniques for Gingival Recession Treatment.
Brief Title: Analysis of Root Coverage Stability.
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: University of Modena and Reggio Emilia (Other); University of Firenze and Siena, Napoli, Italy (Other); The European Research Group on Periodontology (ERGOPerio) (Network)
Responsible Party: Principal Investigator, CARLO BERTOLDI, Professor, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: RB008723
Record Dates: First submitted 2022-06-22; First posted 2022-06-30 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Gingival Recession; Surgery; Oral Disease
Keywords: Gingival recession; Root coverage; Subepithelial tissue graft
MeSH Terms: conditions — Gingival Recession; Mouth Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Langer & Langer technique: Participants undergoing Langer & Langer surgical technique
  Interventions: Procedure: Gingival recession regenerative surgery
- Nelson' modified technique: Participants undergoing Nelson' modified surgical technique
  Interventions: Procedure: Gingival recession regenerative surgery
- Coronally advanced flap and subepithelial graft: Participants undergoing Coronally advanced flap and subepithelial graft surgical technique
  Interventions: Procedure: Gingival recession regenerative surgery

INTERVENTIONS:
Procedure: Gingival recession regenerative surgery — Bilaminar technique was performed by the same trained operator, opening a primary flap in correspondence of the recession site. Tissue was harvested from palatal donor site and grafted beneath the primary flap

SUMMARY:
One-hundred and one healthy participants (221 gingival recessions-GRs) were treated from 1987 to 1996. The probing depth (PD), keratinized tissue width (KTW), gingival recession depth (RD), gingival recession width (RW), gingival recession area (RA) were evaluated and considered at baseline and along time. The obtained data will be evaluated and compared.

DETAILED DESCRIPTION:
Dental-periodontal procedures and clinical measurements.

Dental and periodontal conditions were assessed and treated according to needs in all participants. Emergencies, such as pain or acute dental-periodontal infections, were treated to establish a stable dental-periodontal condition. Cause-related therapy, including patient motivation and professional oral hygiene, was planned and completed.

At the end of cause-related therapy, the following baseline clinical measurements were taken by an investigator: probing depth (PD), keratinized tissue width (KTW), full-mouth plaque scores (FMPS), full-mouth bleeding scores (FMBS), bleeding on probing (BoP), gingival recession depth (RD), gingival recession width (RW), and gingival recession area (RA).

PD and KTW were evaluated using a periodontal probe (University of North Carolina Probe 15 tip) to the nearest 0.5mm. PD was measured at 4 aspects per tooth axially, from the free gingival margin to the most apical part of the sulcus, and, additionally, PD at the mid buccal point; KTW at the mid-buccal point, from the free gingival margin to the mucogingival-junction (MGJ). FMPS was recorded as the percentage of total tooth surfaces (4 aspects per tooth) displaying the presence of plaque, FMBS was calculated as the percentage of total tooth surfaces (4 aspects per tooth) showing bleeding on probing (BoP) was dichotomously assessed.

The bi-dimensional shape of each exposed root surface was reproduced with a lead sheet template. The template had the shape of a triangle with a curved base lining the cemento-enamel-junction (CEJ) and two sides lining the mesial and distal margins of the GR merging at the most apical point of the GR. All templates were measured, coded and stored. The following measurements were recently repeated using an image analysis software: RD, from the most apical point of the triangle to the base; RW, measured at the CEJ level (i.e., at the base of the template) and RA, as the total template area.

These measurements were performed from baseline (before surgery).

Surgery.

All surgical procedures were performed by the same trained operator under local anesthesia.

The recipient site started with an intrasulcular incision on the buccal aspect of the involved teeth. The incision was mesio-distally extended to dissect the buccal aspect of the adjacent papillae. Two oblique releasing incisions were performed from the mesial and distal sides of the horizontal incisions beyond MGJ. A full thickness trapezoid flap, next the dental roots, was raised. Partial dissection was made next the papillae and, apically, at the interproximal places.

After the initial preparation of the recipient site and flap, the bilaminar technique required the withdrawal of palatal connective graft. At the palatal donor site, a horizontal incision was made about 3 mm apical to the free gingival margin. For the epithelial connective tissue graft (ECTG), a second incision was made undermining and splitting the palatal flap. Vertical incisions were carried out mesially and distally joining them to the horizontal incision and performing the palatal flap. Another horizontal incision was made apically on the connective tissue to sever the graft tissue. The graft tissue, 1-1.5 mm thick, was placed in the recipient site to cover the exposed dental roots as far as the CEJ, enlarging mesially and distally on the preserved connective and periosteum of the interproximal sites. Absorbable interrupted and compressive subperiosteal sutures were performed to give stability to the graft. Then, if need to ensure flap mobilization and passivity, a partial thickness dissection was made beyond the MGJ, leaving the underlying periosteum in place and release also the muscle tension, allowing the passive mobilization of the flap that had to cover completely the connective tissue graft (CTG) and the dental roots over the CEJ at least of 2mm. The partial thickness dissection was performed immediately before the graft positioning and suture to avoid flap suffering. The pedicle flap was sutured without residual tension. Each of these surgical techniques could be advantageously used both in cases of single or multiple gingival recessions (GRs).

After surgery, patients were instructed to discontinue toothbrushing of the treated area for 7-10 days. Patients were reinforced to use the roll technique, by soft-bristle toothbrushing outside the treated area during the first month after surgery. Interdental brushes and dental floss in the treated area were forbidden for 1-month. Flap sutures were removed after 7-10 days, and therefore the same toothbrushing prescriptions performed after surgery for outside areas were introduced also in the treated areas. Chlorhexidine rinses were prescribed twice a day for 1 min. About 1-month after surgery, all patients were instructed to resume mechanical tooth cleaning. Patients were recalled for professional supportive care in accordance with Italian health rules and regulations on public dentistry (Essential·Level·of·Assistance - LEA), Law no.·419-30·November·1998, regulating the public dentistry) every 6-24 months whenever possible, and ever in case of need. Patients were recalled for clinical re-evaluations.

ELIGIBILITY:
Inclusion Criteria:

Absence of relevant medical conditions: Medical history of good health. Good oral hygiene: full-mouth plaque score (FMPS) ≤20%. Low level of residual infection: full-mouth bleeding score (FMBS) ≤20%. Participants showing good levels of compliance were selected. Presence of at least one tooth presenting with gingival recession (GR) requiring subepithelial tissue graft, and with identifiable cement-enamel junction (CEJ).

GR exhibiting an identifiable cemento-enamel junction, and absence of plaque or bleeding on probing (BoP) in the sites scheduled for the procedure.

GR defects Miller Class I or II without furcation involvement.

Exclusion Criteria:

Pregnant or lactating. Smokers and participants with history of alcohol abuse. Periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants screened for the presence of at least one tooth presenting with gingival recession requiring subepithelial tissue graft (bilaminar technique), examined and treated from 1987 at the Periodontology Unit of Dentistry and Oral-Maxillofacial Surgery of Modena University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 1987-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Periodontal pocket probing depth (PD) | From surgery to December 2023
  Measurements of the periodontal pocket depth in millimeters
Keratinized tissue width (KTW) | From surgery to December 2023
  Measurements of the width of keratinized tissue (gingiva), in millimeters, from the free gingival margin to the mucogingival junction
Gingival recession depth (RD) | From surgery to December 2023
  Measurements of the depth of the gingival recession, in millimeters, from the cementoenamel junction to the most apical part of the gingival recession
Gingival recession width (RW) | From surgery to December 2023
  Measurements of the width of the gingival recession, in millimeters, from the mesial to distal part of the uncovered cementoenamel junction
Gingival recession area (RA) | From surgery to December 2023
  Measurements of the area, in square millimeters, of the gingival recession

SECONDARY OUTCOMES:
Correlation between initial and late measurements of probing depth (PD) | From surgery to December 2023
  Evaluation of mutual correlation of probing depth (PD) with all the measured indices listed as primary outcome
Correlation between initial and late measurements of keratinized tissue width (KTW) | From surgery to December 2023
  Evaluation of mutual correlation of keratinized tissue width (KTW) with all the measured indices listed as primary outcome
Correlation between initial and late measurements of gingival recession depth (RD) | From surgery to December 2023
  Evaluation of mutual correlation of gingival recession depth (RD) with all the measured indices listed as primary outcome
Correlation between initial and late measurements of gingival recession width (RW) | From surgery to December 2023
  Evaluation of mutual correlation of gingival recession width (RW) with all the measured indices listed as primary outcome
Correlation between initial and late measurements of gingival recession area (RA) | From surgery to December 2023
  Evaluation of mutual correlation of gingival recession area (RA) with all the measured indices listed as primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Bertoldi, MD DDS, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- Periodontology Unit of Dentistry and Oral-Maxillofacial Surgery of the Modena University Hospital, Modena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasperini G, Acunzo R, Pellegrini G, Pagni G, Tonetti M, Pini Prato GP, Cortellini P. Predictor factors for long-term outcomes stability of coronally advanced flap with or without connective tissue graft in the treatment of single maxillary gingival recessions: 9 years results of a randomized controlled clinical trial. J Clin Periodontol. 2018 Sep;45(9):1107-1117. doi: 10.1111/jcpe.12932. Epub 2018 Aug 20. PMID 29777632
- [Background] Chambrone L, Tatakis DN. Long-Term Outcomes of Untreated Buccal Gingival Recessions: A Systematic Review and Meta-Analysis. J Periodontol. 2016 Jul;87(7):796-808. doi: 10.1902/jop.2016.150625. Epub 2016 Feb 15. PMID 26878749
- [Background] Chambrone L, Salinas Ortega MA, Sukekava F, Rotundo R, Kalemaj Z, Buti J, Pini Prato GP. Root coverage procedures for treating localised and multiple recession-type defects. Cochrane Database Syst Rev. 2018 Oct 2;10(10):CD007161. doi: 10.1002/14651858.CD007161.pub3. PMID 30277568
- [Background] Pini-Prato GP, Cairo F, Nieri M, Franceschi D, Rotundo R, Cortellini P. Coronally advanced flap versus connective tissue graft in the treatment of multiple gingival recessions: a split-mouth study with a 5-year follow-up. J Clin Periodontol. 2010 Jul;37(7):644-50. doi: 10.1111/j.1600-051X.2010.01559.x. Epub 2010 May 11. PMID 20492074
- [Background] Pini Prato GP, Franceschi D, Cortellini P, Chambrone L. Long-term evaluation (20 years) of the outcomes of subepithelial connective tissue graft plus coronally advanced flap in the treatment of maxillary single recession-type defects. J Periodontol. 2018 Nov;89(11):1290-1299. doi: 10.1002/JPER.17-0619. Epub 2018 Aug 10. PMID 29873085
- [Background] Francetti L, Weinstein R, Taschieri S, Corbella S. Coronally Advanced Flap With or Without Subepithelial Connective Tissue Graft for the Treatment of Single Recession: 5-Year Outcomes from a Comparative Study. Int J Periodontics Restorative Dent. 2018 November/December;38(6):819-825. doi: 10.11607/prd.3036. Epub 2018 Feb 16. PMID 29451926
- [Background] Carvalho PF, da Silva RC, Cury PR, Joly JC. Modified coronally advanced flap associated with a subepithelial connective tissue graft for the treatment of adjacent multiple gingival recessions. J Periodontol. 2006 Nov;77(11):1901-6. doi: 10.1902/jop.2006.050450. PMID 17076617
- [Background] Leknes KN, Amarante ES, Price DE, Boe OE, Skavland RJ, Lie T. Coronally positioned flap procedures with or without a biodegradable membrane in the treatment of human gingival recession. A 6-year follow-up study. J Clin Periodontol. 2005 May;32(5):518-29. doi: 10.1111/j.1600-051X.2005.00706.x. PMID 15842269
- [Background] Nickles K, Ratka-Kruger P, Neukranz E, Raetzke P, Eickholz P. Ten-year results after connective tissue grafts and guided tissue regeneration for root coverage. J Periodontol. 2010 Jun;81(6):827-36. doi: 10.1902/jop.2010.090632. PMID 20450359
- [Background] Kuis D, Sciran I, Lajnert V, Snjaric D, Prpic J, Pezelj-Ribaric S, Bosnjak A. Coronally advanced flap alone or with connective tissue graft in the treatment of single gingival recession defects: a long-term randomized clinical trial. J Periodontol. 2013 Nov;84(11):1576-85. doi: 10.1902/jop.2013.120451. Epub 2013 Feb 22. PMID 23432657
- [Background] Zucchelli G, Mounssif I, Mazzotti C, Stefanini M, Marzadori M, Petracci E, Montebugnoli L. Coronally advanced flap with and without connective tissue graft for the treatment of multiple gingival recessions: a comparative short- and long-term controlled randomized clinical trial. J Clin Periodontol. 2014 Apr;41(4):396-403. doi: 10.1111/jcpe.12224. Epub 2014 Jan 22. PMID 24382170
- [Background] Jepsen K, Stefanini M, Sanz M, Zucchelli G, Jepsen S. Long-Term Stability of Root Coverage by Coronally Advanced Flap Procedures. J Periodontol. 2017 Jul;88(7):626-633. doi: 10.1902/jop.2017.160767. Epub 2017 Mar 17. PMID 28304210
- [Result] Barootchi S, Tavelli L, Di Gianfilippo R, Byun HY, Oh TJ, Barbato L, Cairo F, Wang HL. Long term assessment of root coverage stability using connective tissue graft with or without an epithelial collar for gingival recession treatment. A 12-year follow-up from a randomized clinical trial. J Clin Periodontol. 2019 Nov;46(11):1124-1133. doi: 10.1111/jcpe.13187. Epub 2019 Sep 9. PMID 31446625
- [Derived] Bertoldi C, Consolo U, Lalla M, Zaffe D, Tanza D, Cairo F, Cortellini P. Long-term stability (21-30 years) of root coverage outcomes using sub-epithelial connective tissue grafts at single or multiple gingival recessions: A longitudinal case series. J Clin Periodontol. 2024 Jan;51(1):2-13. doi: 10.1111/jcpe.13882. Epub 2023 Oct 5. PMID 37794814